CLINICAL TRIAL: NCT03637595
Title: Efficacy and Mechanisms of Energy Medicine to Decrease Chronic Knee Pain in Outpatient Settings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study lapsed due to COVID-19.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 18-00600
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Ostheoporosis of the Knee
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive Control Group (Active Comparator): Acupuncture
  Interventions: Procedure: Acupuncture
- Negative Control Group (Sham Comparator): Sham Intervention
  Interventions: Procedure: Sham Energy Medicine
- Energy Medicine (EM) Intervention (Experimental): Energy Medicine by an energy medicine practitioner
  Interventions: Procedure: Enery Medicine Intervention

INTERVENTIONS:
Procedure: Acupuncture — 3 sessions of acupuncture will be the reference therapy against which the energy medicine intervention is being compared.
  Arms: Positive Control Group
Procedure: Enery Medicine Intervention — 3 sessions performed by Energy Medicine practitioner, who will perform an assessment followed by the intervention.
  Arms: Energy Medicine (EM) Intervention
Procedure: Sham Energy Medicine — a non-energy trained confederate to be determined from the clinical research coordinators and non traditional volunteers enrolled administering assessments and providing therapeutic company.
  Arms: Negative Control Group

SUMMARY:
This study will assess the efficacy and mechanisms behind Energy Medicine in reducing chronic knee pain within an outpatient setting. This study will investigate a form of Energy Medicine (EM) performed by a natural solo practitioner, using a standard number of three sessions, which will compare to both positive and negative control groups. The positive control group will receive acupuncture and the negative control group will receive a sham intervention.

ELIGIBILITY:
Inclusion Criteria:

* Presence of knee pain lasting for at least six months
* No radiation of knee pain
* No acupuncture treatments in the previous six months
* Failure to respond completely to the medications given by their orthopedic or pain management specialist
* Knee pain on most days (4 out of 7 days of the week) with average self-reported severity of 4 or more out of 10 on a numeric rating scale (NRS)
* Complaints of morning stiffness lasting less than 30 minutes
* Not be in active physical therapy (PT) for the duration of the trial.
* Adult patients ≥18 years of age
* English speaking

Exclusion Criteria:

* Any concurrent diagnosis of systemic disease
* Other concurrent treatments such as massage, Acupcunture, PT or any kind of Energy Medicine
* Bleeding disorder
* Trypanophobia (fear of needles or injections).
* Have medical condition that causes difficulty in saliva production/collection (i.e.: Sjogren's Syndrome)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Pain Level measured by 11- Point Numeric Rating Scale (NRS) | 18 Months
  11 point scale (0-10) asking patient leve of discomfort. A state of no pain is "0" and worst pain is "10"
Pain Level measured by Visual Analog Scale (VAS) | 18 Months
  used for quantification of pain; psychometric response scales used to measure subjective characteristics or attitudes and have been used in the past for a multitude of disorders, as well as in market research and social science investigations, among others
Self Reported Physical Function measured y the Western Ontario and McMaster Universities Ostheoarthritic Index (WOMAC) | 18 Months
  self-administered questionnaire consisting of 24 items divided into 3 subscales:[1]
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Siminovich-blok, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Requests should be directed to siminb01@nyumc.org To gain access, data requestors will need to sign a data access agreement.